CLINICAL TRIAL: NCT03760991
Title: A Multicenter, Multinational, Prospective, Interventional, Single-arm, Phase IV Study Evaluating the Clinical Efficacy and Safety of 26 Weeks of Treatment With Insulin Glargine 300 U/mL (Gla-300) in Patients With Type 2 Diabetes Mellitus Uncontrolled on Basal Insulin
Brief Title: Evaluation of the Efficacy and Safety of Insulin Glargine 300 U/mL in Patients With Type 2 Diabetes Mellitus Uncontrolled on Other Kinds of Insulin
Acronym: ARTEMIS-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS15396; U1111-1203-8663 (Other: UTN)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insulin glargine (U300) (Experimental): Insulin glargine (U300) (Gla-300) once daily for 26 weeks on top of any other antidiabetic treatment except other basal insulin
  Interventions: Drug: INSULIN GLARGINE (U300)

INTERVENTIONS:
Drug: INSULIN GLARGINE (U300) — Pharmaceutical form: Solution for injection in a prefilled pen
  Route of administration: Subcutaneous
  Other Names: HOE901, Toujeo, Gla-300

SUMMARY:
Primary Objective:

To assess the efficacy of Gla-300 on glycemic control measured by hemoglobin A1c (HbA1c) change in patients with type 2 diabetes mellitus (T2DM) uncontrolled with their current basal insulin following the switch to Gla-300.

Secondary Objectives:

To evaluate the effects of Gla-300 on glycemic control, treatment satisfaction, and health care resource utilization (HCRU) outcomes.

To evaluate the safety of Gla-300.

DETAILED DESCRIPTION:
Study duration per participant is approximately 29 weeks including a screening period of up to 2 weeks, a 26-week treatment period, and a post treatment follow-up phone call visit at Week 27.

ELIGIBILITY:
Inclusion criteria :

* Participants with type 2 diabetes mellitus.
* Participants on "standard of care" basal insulin therapy administered once or twice daily, as per labeling for at least 6 months prior to screening visit, with or without other antidiabetics approved for using with insulin.
* Glycated hemoglobin (HbA1c) between 7.5% (58 mmol/mol) and 10% (86 mmol/mol) inclusive, during screening.
* Fasting plasma glucose values above 130 mg/dL.

Exclusion criteria:

* Unstable basal insulin regimen in the last 8 weeks prior to screening visit (ie, type of insulin and time/frequency of the injection, insulin doses [variation more than ±20%]).
* Treatment with insulin other than basal insulin: mixed insulin (premixes), rapid insulin, fast acting insulin analogues in the last 6 months before screening visit (use ≤10 days in relation to hospitalization or an acute illness is accepted).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) | Baseline to Week 26
  Absolute change in HbA1c

SECONDARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) | Baseline to Week 12
  Absolute change in HbA1c
Participants with HbA1c below 7% | Week 12 and 26
  Percentage of participants with HbA1c below 7%
Participants with fasting self-monitored plasma glucose (SMPG) of 80 to 110 mg/dL (4.4 to 7.2 mmol/L) | Week 12 and 26
  Percentage of participants reaching targeted fasting SMPG of 80 to 110 mg/dL (4.4 to 7.2 mmol/L)
Change in fasting SMPG | Baseline to Week 26
  Absolute change in fasting SMPG
Change in SMPG profile | Baseline to Week 26
  Absolute change in SMPG profile
Change in fasting plasma glucose (FPG) | Baseline to Week 26
  Absolute change in FPG
Percentage of participants requiring rescue therapy | Baseline to Week 12 and 26
  Percentage of participants requiring rescue therapy by additional antidiabetic medication
Number of participants with hypoglycemia events | Baseline to Week 26
  Number of participants with at least 1 hypoglycemia event
Number of participants with adverse events (AEs) | Baseline to Week 27
  Number of participants with AEs, serious adverse events (SAEs) (including hypoglycemic episodes associated with seizures, coma, or unconsciousness).
Change in Treatment satisfaction | Baseline to Week 26
  Change in treatment satisfaction as measured by insulin treatment satisfaction questionnaire
Number of participants with health care utilization | Baseline to Week 26
  Number of participants with health care utilization, including hospitalization, emergency room visits, and office [or specialty] visits

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- Investigational site Argentina, Buenos Aires, Argentina
- investigational site COLOMBIA, Colombia, Colombia
- investigational site Egypt, Egypt, Egypt
- investigational site HONG KONG, Hong Kong, Hong Kong
- investigational site INDIA, India, India
- Investigational site Indonesia, Indonesia, Indonesia
- investigational site LEBANON, Lebanon, Lebanon
- Investigational site Malaysia, Putrajaya, Malaysia
- Investigational site PERU, Hacienda Perú, Peru
- investigational site PHILIPPINES, Philippines, Philippines
- Investigational site Saudi Arabia, Saudi Arabia, Saudi Arabia
- Investigational site South Africa, South Africa, South Africa
- Investigational site Thailand, Thailand, Thailand
- investigational site TURKEY, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Sethi B, Al-Rubeaan K, Unubol M, Mabunay MA, Berthou B, Pilorget V, Vethakkan SR, Frechtel G. Efficacy and Safety of Insulin Glargine 300 U/mL in People with Type 2 Diabetes Uncontrolled on Basal Insulin: The 26-Week Interventional, Single-Arm ARTEMIS-DM Study. Diabetes Ther. 2022 Jul;13(7):1395-1408. doi: 10.1007/s13300-022-01271-7. Epub 2022 Jun 17. PMID 35713873